CLINICAL TRIAL: NCT06378372
Title: Effect of Musical Intervention Based on Piano Learning on Alzheimer's Patients in León (España).
Brief Title: How Does Pianistic Musical Training Influence the Development of Alzheimer's Disease?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Franco Castellanos (Other)
Collaborators: Jesús Ángel Seco Calvo (Unknown); Javier Tejada Garcia (Unknown)
Responsible Party: Sponsor-Investigator, David Franco Castellanos, Assistant professor, Universidad de León
Organization: Universidad de León (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ETICA-ULE-064-2023
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Dementia of Alzheimer Type; Dementia; Dementia, Vascular; Dementia, Mixed; Dementia Frontal; Dementia With Lewy Bodies; Cognitive Decline; Neurologic Disorder; Neurologic Dysfunction; Neurologic Deficits
Keywords: Alzheimer; Neuropsicology; Music; Piano; Rehabilitación; Music Theraphy
MeSH Terms: conditions — Dementia; Dementia, Vascular; Mixed Dementias; Lewy Body Disease; Cognitive Dysfunction; Nervous System Diseases; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: An intervention based on teaching the piano in an individualized way
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Grupo 0 (Experimental): Group on which the pianistic intervention will be carried out
  Interventions: Behavioral: Music therapy based on piano learning

INTERVENTIONS:
Behavioral: Music therapy based on piano learning — The intervention will consist of pianistic training. Patients will receive piano classes adapted to their competence designed to achieve motor, sensory and behavioral control.

SUMMARY:
The goal of this clinical trial is to learn about and describe how pianistic training influences the development of Alzheimer's disease.

The key question is: Can pianistic practice influence the development of Alzheimer's disease?

Participants will receive piano lessons for 4 weeks (20 sessions) and we will evaluate the evolution of the different parameters described by the tests carried out.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a chronic neurodegenerative disease that affects different areas of the brain causing progressive changes in behavior, memory loss, decreased personal autonomy and various cognitive alterations. (Masters et al., NINDS, 2019; Alzheimer's Association, 2020)

According to the World Health Organization (WHO), currently around 50 million people suffer from some type of diagnosed dementia, of which 60-70% of them report some type or degree of EA. (Alzheimer's Association, 2020; WHO, 2020)

Not only is AD considered a worrying pathology today, but the forecast for medium and long term envisions a severe evolution that will reach 75 million cases in 2030 and 132 million in 2050. (Scheltens et al., 2016; MSCBS, 2019) Specifically in Spain there are more than 700,000 patients currently diagnosed and the forecast is that this number of people affected by AD will double in 2050. (MSCBS, 2019)

Since at the beginning of the s. XX the characteristics of AD were described for the first time (Mauer. K, 2006), scientific research has been, in its beginnings, aimed at alleviating the disease since a pharmacological point of view with modestly effective results (López, 2015) and effects secondary, sometimes unwanted. It therefore seems necessary to address the research and treatment of this disease from a non-pharmacological prism in which music has shown a high degree of efficiency with no adverse effects.

It is at this point that other alternative therapies such as music therapy take center stage. providing notable evidence of the brain activation that occurs, especially when the patient receives sound stimuli. (Peretz, 2005)

The value of music is evident in the numerous cases of musicians (pianists, violinists...) who after a diagnosis of AD begin to experience cognitive and physical deterioration expected, however, this degenerative process does not seem to affect their motor or intellectual to play his instrument even when the disease is in its most severe stage. (Pladdy, 2011)

Thus arises the need to go deeper and discover how music "interferes" in the process. neurodegenerative caused by AD and how it can partner with the patient to, potentially improve your quality of life, strengthen your cognitive reserve, become a useful routine and viable to implement active aging and, ultimately, accompany the patient during evolution of this pathology and, why not?, when the time comes to reverse its advance.

The most common interventions that focus on music as a vehicle to treat AD are aimed at mitigating stress, reducing anxiety and controlling agitation through listening, dancing or singing. (Baird, 2009) However, there are no studies that describe the influence that has to learn to play a musical instrument, in the case of this doctoral thesis: the piano, in the evolution of AD.

The piano is an instrument capable of mobilizing sight, hearing, touch, gross and fine motor skills, perception and emotion activating and making multiple parts of the brain interact (Paxinos, 2004) (hippocampus, cerebral cortex) which, judging by the latest studies, are related to the detection, evolution and treatment of AD.

Hypothesis:

- A therapy based on teaching patients with AD to play the piano may be beneficial for increase your Cognitive Reserve Capacity and improve your Quality of Life.

In this sense, it has been shown that complex mental activity throughout the life cycle can work as a neuroprotective factor in AD. (Valenzuela, 2006)

General objective:

- Analyze the effects of a musical intervention based on piano learning on Alzheimer's patients in León.

Specific objectives:

* Generate a specific didactic program adapted to Alzheimer's patients based on in acquiring piano skills.
* Involve the members under study in a prolonged musical experience in time (4 weeks) and value its significance from a therapeutic point of view.
* Evaluate the evolution of the acquisition of sensory and musical skills in the course of the intervention.
* Carry out a longitudinal-correlational study of the results obtained pre-post intervention. (Spss)
* Make an evaluation of the didactic programming and the quality and suitability of the intervention at the end of it to, where appropriate, modify and reorient the aspects susceptible to improvement.

Methodology

The preparation of this study will be structured around three phases. A first phase of documentation on the state of the matter and preparation of the teaching materials that will form part of the resources necessary to carry out the therapeutic intervention. A second phase that will consist of the intervention itself, as well as the collection of the data provided by the control of the different variables subject to study, and finally, a third phase consisting of the evaluation of the data collected, as well as a critical assessment of the pedagogical procedure and, in If applicable, a proposal for an improvement plan for this intervention will be made.

The general methodology of the musical intervention will be an active, participatory, inclusive methodology and integrative, based on project-based learning. It will take into account at all times the uniqueness of each patient, therefore applying personalized attention. In it they will be used musical and extra-musical resources as formative elements, also valuing the Free improvisation as an artistic formula and musical and emotional expression.

The didactic programming will be aimed at developing motor control, developing the connection. Be careful, listen, and will also try to develop the capacity for self-criticism and frustration management, anxiety and emotional control.

The specific methodology of each therapy session will be defined in each of the units that they will make up the didactic programming prepared to carry out the intervention. Having in keep in mind that each session will last 30 minutes, the general methodological dynamic will revolve around this temporary organization:

Activation: 5´Making contact with himspace - teacher - instrument. Development: 20´ Pedagogical intervention. Relaxation: 5´Back to the calm.

Tests and variables:

Age, sex, socio-economic-cultural profile, nutritional status, motor status and other clinical data ofpatient interest. (tension, glucose...)

Cognitive state: (Minimal + (clock, cancellation and Ways))

* Global
* Domains: Memory (procedural and declarative. Language, Visuospatial.

Attention.

Visoconstructive, Executive abilities. Behavioral status: (medication) Typology of dementia (inclusion and exclusion criteria in the study) Degree of AD: (Mild moderate, severe, very severe) State of global deterioration.

Functional tests (RDRS-2 Rapid Disability Assessment Scale)

Cognitive evaluation tests: MOCA, WAIS-IV (digits), IST, ZAZZO, Trail Making Test, Clock, Fluency Verbal/categorical.

Neuropsychiatric evaluation test:

* Behavioral disorders: BEHAVE-AD (Sclan 1996)
* Frequency and severity of symptoms: Neuropsychiatric Inventory (NPI) (Cummings, 1994):
* NPI-Q gravity part
* NPI-Q caregiver stress
* Evaluation of the severity of the disease (CDS and GDR Scales)
* Evaluation of the caregiver's burden (Zarit test)

MEDIA AND MATERIAL RESOURCES AVAILABLE

This Initial Research Plan will be presented to the management of ALZHEIMER LEON to make a joint assessment of the suitability and viability of the proposed intervention.

Once approved its execution, the subjects who will make up the sample on which it will be determined will be determined. Will enhance the intervention. A series of tests will be carried out to determine the characteristics of the itself and inclusion/exclusion criteria will be set according to the needs of the study.

Additionally, there will be the departments of interest for the study (Psychology, psychiatry, therapists, social workers...) In addition, this intervention project will be presented to different entities to achieve maximum economic, human and institutional coverage. In this sense, some have been tested private and public institutions such as the Valverde de La Virgen School of Music through its City Council or JJMM-ULE, all of them showing great interest in the study and valuing positively their participation in the research without limiting for the moment the role that each of them they would take in the process.

To carry out the intervention it will be necessary to have a specialist pianist teacher, with a solid musical and pedagogical training and with an additional approach to the particularities of the sample and dynamics of the didactic programming prepared for the study. It will be very important and It is also necessary to have adequate financing to meet the expenses derived from the hiring and training of this professional and other unexpected expenses.

At all times we will try to find appropriate synergies with other entities interested in this study to join forces that give economic viability and dissemination to the project and its results through agreements, collaborations, donations or contributions of any nature.

ELIGIBILITY:
Inclusion Criteria:

- Patients in State of global deterioration Levels GDS 2 3 and 4.

Exclusion Criteria:

* Other patients in GDS groups (not 2, 3 and 4)
* The selected subject does not cooperate during intervention.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
State of global deterioration | Pre-intervention, Post-intervention (after four weeks of intervention), Follow up after 6 month intervention.
  GDS 1 - 7
Minimental Test | Pre-intervention, Post-intervention (after four weeks of intervention), Follow up after 6 month intervention.
  0-24
RDRS-2 Rapid Disability Assessment Scale | Pre-intervention, Post-intervention (after four weeks of intervention), Follow up after 6 month intervention.
  18-72
MONTREAL COGNITIVE ASSESSMENT (MOCA) | Pre-intervention, Post-intervention (after four weeks of intervention), Follow up after 6 month intervention.
  0-30
WAIS-IV | Pre-intervention, Post-intervention (after four weeks of intervention), Follow up after 6 month intervention.
  0-160
Behavioral disorders: BEHAVE-AD | Pre-intervention, Post-intervention (after four weeks of intervention), Follow up after 6 month intervention.
NPI - CUMMINGS | Pre-intervention, Post-intervention (after four weeks of intervention), Follow up after 6 month intervention.
  0-120
Evaluation of the caregiver's burden (Zarit test) | Pre-intervention, Post-intervention (after four weeks of intervention), Follow up after 6 month intervention.
  0-88

CONTACTS AND LOCATIONS:
Overall Officials: David Franco-Castellanos, Sr, Principal Investigator — Universidad de León
Locations (1):
- Universidad de León, León, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzheimer´s Association. (2020). 2020 Alzheimer´s Disease Facts and Figures. Alzheimer´s & Dementia: The Journal of the Alzheimer Association, 16(3), 391-460. Doi: 10.1002/alz.12068
- [Background] Baird A, Samson S. Memory for music in Alzheimer's disease: unforgettable? Neuropsychol Rev. 2009 Mar;19(1):85-101. doi: 10.1007/s11065-009-9085-2. Epub 2009 Feb 13. PMID 19214750
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Hanna-Pladdy B, MacKay A. The relation between instrumental musical activity and cognitive aging. Neuropsychology. 2011 May;25(3):378-86. doi: 10.1037/a0021895. PMID 21463047
- [Background] López O, Tratamiento farmacológico de la enfermedad de Alzheimer y otras demencias. (2015) Recuperado de: http://www.scielo.edu.uy/scielo.php?pid=S1688-423X2015000200003&script=sci_arttext&tlng=pt
- [Background] Maurer K, Maurer U. Alzheimer. La vida de un médico, la historia de una enfermedad. Madrid: Díaz de Santos; 2006.
- [Background] MSCBS. Ministerio de Sanidad, Consumo y Bienestar Social (2019) Plan integral de Alzheimer y otras Demencias (2019-2023) Recuperado de: https://mscbs.gob.es/profesionales/saludPublica/docs/Plan_Integral_Alzheimer_Octubre_2019.pdf
- [Background] NINDS. National Institute of Neurological Disorders and Stroke. (2019). Recuperado de: https://www.ninds.nih.gov/Disorders/All-Disorders/Alzheimers-Disease Information-Page
- [Background] Paxinos, G. y Mai, J. (2004). The human nervous system. Academic Press, Inc.
- [Background] Peretz I, Zatorre RJ. Brain organization for music processing. Annu Rev Psychol. 2005;56:89-114. doi: 10.1146/annurev.psych.56.091103.070225. PMID 15709930
- [Background] Sclan S, Saillon A, Franssen E, et al. The behavior pathology in Alzheimer's disease ratings scale (BEHAVE-AD): reability and analisys of symptom category scores. Int J Geriatr Psychiatry, 1996; 11: 819-830.
- [Background] Scheltens P, Blennow K, Breteler MM, de Strooper B, Frisoni GB, Salloway S, Van der Flier WM. Alzheimer's disease. Lancet. 2016 Jul 30;388(10043):505-17. doi: 10.1016/S0140-6736(15)01124-1. Epub 2016 Feb 24. PMID 26921134
- [Background] Sultzer DL, Levin HS, Mahler ME, High WM, Cummings JL. Assessment of cognitive, psychiatric, and behavioral disturbances in patients with dementia: the Neurobehavioral Rating Scale. J Am Geriatr Soc. 1992 Jun;40(6):549-55. doi: 10.1111/j.1532-5415.1992.tb02101.x. PMID 1587970
- [Background] Tariot PN, Mack JL, Patterson MB, Edland SD, Weiner MF, Fillenbaum G, Blazina L, Teri L, Rubin E, Mortimer JA, et al. The Behavior Rating Scale for Dementia of the Consortium to Establish a Registry for Alzheimer's Disease. The Behavioral Pathology Committee of the Consortium to Establish a Registry for Alzheimer's Disease. Am J Psychiatry. 1995 Sep;152(9):1349-57. doi: 10.1176/ajp.152.9.1349. PMID 7653692
- [Background] Valenzuela MJ, Sachdev P. Brain reserve and dementia: a systematic review. Psychol Med. 2006 Apr;36(4):441-54. doi: 10.1017/S0033291705006264. Epub 2005 Oct 6. PMID 16207391